CLINICAL TRIAL: NCT01200615
Title: The Nocebo Effect: a Prospective Study of Informed Consent as a Factor in the Prevalence of SSRI's Side Effects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Dr. Uri Nitzan, Shalvata Mental Health Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 025622648
Record Dates: First submitted 2010-08-26; First posted 2010-09-13 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Depression
Keywords: nocebo side-effects SSRI informed consent
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Explanation about common side effects (Other): 50 patients started on SSRI's will be updated about its common side effects
  Interventions: Behavioral: Wording of the explenation on side-effects as part of the informed consent.
- Explaning side effects and the nocebo effect (Other): subjects started on SSRI's will be updated about its common side effects and the nocebo effect
  Interventions: Behavioral: Wording of the explenation on side-effects as part of the informed consent.
- explanation about the nocebo effect (Other): 3. 50 patients started on SSRI's will receive an explenation on the nocebo effect, but will not be updated about common side-effects. Nonetheless, they will be informed of severe side-effects.
  Interventions: Behavioral: Wording of the explenation on side-effects as part of the informed consent.

INTERVENTIONS:
Behavioral: Wording of the explenation on side-effects as part of the informed consent. — Subjects will hear different versions of the description of SSRI's side-effects and the nocebo effect.

SUMMARY:
In this study we invetigate the influence of the nocebo effect (as part of obtaining informed consent) on the prevalence of side-effects. The study is prospective, focusing on the connection between what the physicians says to the patient about side-effects to the frequency of these side effects during treatment period. We also inquire whether informing the patient about the existence of the nocebo effect influences the extent of phenomena.

DETAILED DESCRIPTION:
In this study the investigators wish to inquire whether the nature of the explenation given to the patient as part of informed consent has an effect on the prevalence of side-effects. The study will take place in the out-patient clinic at the Shalvata Mental health Center. Three arms are included:

1. 50 patients started on SSRI's will be updated about its common side effects
2. 50 patients started on SSRI's will be updated about its common side effects and will receive an explenation on the nocebo effect
3. 50 patients started on SSRI's will receive an explenation on the nocebo effect, but will not be updated about common side-effects. Nonetheless, they will be informed of severe side-effects.

Following the prescription of an SSRI the subjects will we enter the follow-up phase of the study. They will attend two follow-up meetings: 3 days after the initiation point and one month after the starting point. During each meeting they will be asked to fill the Antidepressant Side-Effect Checklist (ASEC)and the General Health Questionnaire (GHQ).

ELIGIBILITY:
Inclusion Criteria:

1. age 18-60
2. started on an SSRI

Exclusion Criteria:

* Psychotic spectrum disorder
* Suicidality
* Sensitivity to SSRI
* Has taken the prescribed SSRI in the past

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
The prevalence of side-effects | 6 weeks
  We are interested in the possible influence of the physicians wording upon recieving informed consend from the patient and the prevalence of side-effects

CONTACTS AND LOCATIONS:
Overall Officials: Uri Nitzan, MD, Principal Investigator — Shalvata Mental Health Center
Locations (1):
- Shalvata Mental Health Center, Hod HaSharon, Israel